2017年11日

## **Case Report Form**

A Prospective, Double-Blind, Randomized,
Placebo-Controlled, Parallel-Group,
Proof-of-Concept Study to Investigate the Effect
Effectiveness of KEFPEP® on Regulating Blood
Pressure

Protocol No.: PHP1705H01

Screen No.: S \_\_\_ \_\_

Subject Initials: \_\_\_ \_\_

CRF Version: 1.0

Date: Jul-12-2017

| Screen No. | Subject Initials | Screening<br>Visit 1 |
|---|---|---|
| Date of visit:/ / | (dd/mmm/yyyy) | |
| Inform | ned Consent Signe | ed and an arrangement |
| Informed consent was given for the parture, scope and possible conseque consent in an understandable manner. | ences of the study were | e explained to the person giving |
| IMPORTANT: Informed consent mo<br>procedures are started. | ust be obtained from | the patient BEFORE any trial |
| Date of informed consent signed: | ! | (dd/mmm/yyyy) |
| | Demographics | |
| Date of birth:/// | (dd/mmm/yyyy) | |
| Gender: Male Female | | |
| Race: | please specify | |
| Height: cm Weig | ht: kg | BMI: kg/ m <sup>2</sup> |
| Smoking habit: Yes No | | |
| Alcohol abuse*: Yes No | | |
| *: Alcohol abuse is classified as ≥ 8 units of participation. The patient with alcohol abuse | | |
| parsopation in patient with accept abuse | anoula de excluded nom a | ic study. |
| F | Pregnancy Test | |
| Is pregnancy test Yes performed: | | |
| No, reason: | ∐ Male | Postmenopause |
| | Hysterectomy | Bilateral tubal Ligation |
| | Other, please sp | |
| Date of assessment:/ | (dd/mmm | /yyyy)<br> |
| Result: Positive Negative | | |

| | Medical History | |
|---|---|---|
| *: Record med | Is there any significant medical history*: Yes No * Record medical histories in the past 6 months prior to Screening visit/ICF date, while specific events (milk allergy and lactose intolerance) prior to Screening visit should be checked without time limitation. | |
| No. | Medical history | Past or Active |
| H | | Past Active |
| H | | Past Active |
| H | | Past Active |
| H | | Past Active |
| H | | Past Active |
| H | | Past Active |
| H | | Past Active |
| н | | Past Active |
| H | | Past Active |
| | ls this the last page ા | used? Yes No |

| Screen No. | Subject Initials | Screening |
|------------|------------------|-----------|

| | Ph | ysical Exa | minations | |
|---|---|---|---|---|
| ls t | Is the examination performed: Yes No | | | |
| Dat | Date of examination:/(dd/mmm/yyyy) | | | |
| | 8:410 | Result | | Specify if abnormal or |
| | Sites/System | Normal | Abnormal | not done |
| 1 | General appearance | | | |
| 2 | Head/ears/eyes/nose/throat | | | |
| 3 | Mouth | | | |
| 4 | Skin | | | |
| 5 | Neck (including thyroid) | | | |
| 6 | Lymph nodes | | en e e e e e e e e e e e e e e e e e e | |
| 7 | Spine | | | |
| 8 | Cardiovascular system | | | |
| 9 | Respiratory system | | | |
| 10 | Gastro-intestinal system | | | |
| 11 | Nervous system | | | |
| 12 | Musculoskeletal system | | | |
| 13 | Blood and blood forming organs | | | |
| 14 | Mental status | | | |
| 15 | Other, specify: | | | |

| Screen No. | Subject Initia | lls | Screening<br>Visit 1 |
|---|---|---|---|
| | Vital Signs | | |
| Is the assessment performed: | Yes No | | |
| Date of assessment:/ | /(dd/mm | m/yyyy) | |
| Body temperature:°C | | | |
| Pulse rate: bpm | | | |
| Respiratory rate: times/ | minute | | |
| Is the assessment performed*: * the subject's office BP will be measu | red at an air-conditioned roo | | ninutes of rest in the |
| sitting position using an electronic sphys Date of assessment:/ | | ım/yyyy) | |
| Systolic Blood Pressure <sup>\$</sup> : Right \$: The arm with higher SBP value will be | arm: mmHg | Left arm: | mmHg |
| Diastolic Blood Pressure: Right | arm: mmHg | Left arm: | <u></u> mmHg |
| | | | 1000 |
| Ele | ectrocardiogram (E0 | CG) | |
| Is the examination performed: | Yes No | | |
| Date of examination:/ | / (dd/mm | nm/yyyy) | |
| Result: Normal Abnorm | al, NCS 🔲 Abnormal, | cs | |
| Abnormal Findings: | | | · |

| Screen No. | Subject Initials | Screening |
|------------|------------------|-----------|

| | | Biochemistry Tests | | |
|---|---|---|---|---|
| ls t | he test performed: Yes | No | | |
| Dat | te of sample:/ | _/ (dd/mmm/yyy | y) | |
| | | | Result | |
| | Item | Value | Normal | Abnormal |
| 1 | Total bilirubin | | | □cs □ncs |
| 2 | Aspartate transaminase (AST) | | | □cs □ncs |
| 3 | Alanine transaminase (ALT) | | | □cs □ncs |
| 4 | Alkaline phosphatase<br>(ALP) | | | ☐cs ☐ncs |
| 5 | Serum creatinine | | | □cs □ncs |
| 6 | Blood urea nitrogen<br>(BUN) | | | □cs □ncs |
| 7 | Uric acid | | | ☐cs ☐ncs |
| 8 | Triglyceride (TG) | | | ☐cs ☐ncs |
| 9 | Total cholesterol (T-Cho) | | | ☐cs ☐ncs |
| 10 | HDL-cholesterol (HDL-C) | | | ☐cs ☐ncs |
| 11 | LDL-cholesterol (LDL-C) | | | □cs □ncs |
| 12 | Glucose (A.C.) | | | □cs □ncs |
| 13 | Hba1c | | | □cs □ncs |
| 14 | Sodium (Na) | | | □cs □ncs |
| 15 | Potassium (K) | | | □cs □ncs |
| 16 | Chloride (CI) | is again | | ☐cs ☐ncs |

| <u>,, </u> | | | | |
|---|---|---|---|---|
| | | Hematology Test | S | |
| ls th | ne test performed: | Yes No | | |
| Dat | e of sample:/ | / (dd/mmm/y | уууу) | |
| | | Malua | | Result |
| | Item | Value | Normal | Abnormal |
| 1 | Hemoglobin | | | ☐cs ☐ncs |
| 2 | Platelet | | | ☐cs ☐ncs |
| 3 | RBC | | | □cs □ncs |
| 4 | WBC | | | □cs □ncs |
| 5 | Neurophils | | | □cs □ncs |
| 6 | Eosinophils | | | ☐cs ☐ncs |
| 7_ | Lymphocyte | | | □cs □ncs |
| .8 | Monocytes | | | □ CS □ NCS |
| 9 | Basophils | | | ☐cs ☐ncs |
| | | and the second s | | *. |
| | | Urinalysis Tests | <b>.</b> | · . |
| ls t | he test performed: | Yes No | | |
| Da | te of sample:/ | /(dd/mmm/ | ′уууу) | |
| | | | | Result |
| | ltem | Value | Normal | Abnormal |
| 1 | WBC | | | ☐cs ☐ncs |
| 2 | RBC | | | ☐cs ☐ncs |
| 3 | PH | | | ☐cs ☐ncs |
| 4 | PROTEIN | | | ☐cs ☐ncs |
| 5 | SUGAR | | | □cs □ncs |

| Screen No. | Subject Initials | Screening<br>Visit 1 |
|------------|------------------|----------------------|

| | Inclusion Criteria | | |
|---|---|---|---|
| | | Yes | No |
| 1 | Male or female patient ages 20 years or older. | | |
| 2 | Belong to either one of the following categories based on JNC 7 as measured by office BP at Screening visit: ➤ Prehypertension (SBP 120 – 139 mmHg or DBP 80 – 89 mmHg) ➤ Stage I hypertension (SBP 140 – 159 mmHg or DBP 90 – 99 mmHg) | | |
| 3 | Body weight $\leq$ 90 kg, and BMI $\geq$ 18.5 kg/m <sup>2</sup> or $<$ 30 kg/m <sup>2</sup> . | | |
| 4 | NOT on any antihypertensive treatment at the time of entry into the study. | | |
| 5 | Willing to comply with the study procedures and follow-ups. | | |
| 6 | A good understanding of the nature of the study and placed signature on the informed consent form. | | |
| | Exclusion Criteria | | |
| 1 | Patients with any of the following conditions within 6 months prior to study participation: > Secondary hypertension > Uncontrolled diabetes mellitus > Renal disease based on the investigator's judgment > Severe hepatic disease with Child-Pugh class C > Severe anaemia > Any malignant disease or serious disease | | |
| 2 | Patients with clinically significant abnormalities in the following laboratory parameters within 2 weeks prior to Screening visit or during the screening period: > HbA1c > 9% > AST or ALT ≥ 3*upper limit of normal (ULN) > Estimated glomerular filtration rate (eGFR) < 50 ml/min/1.73 m² > Serum creatinine ≥ 3*ULN > Hemoglobin < 10 g/dL | | |
| 3 | History of milk allergy and/or lactose intolerance. | | |
| 4 | Alcohol abuse classified as ≥ 8 units of alcoholic consumption per week within 1 month prior to study participation. | | |
| 5 | Constant use of oral medication or supplements affecting blood pressure. | | |
| 6 | Female patients who are pregnant, planning to become pregnant, or lactating. | | |
| 7 | Male or female patients of child-bearing potential do not agree to use an effective method of contraception during the study period. | | |
| 8 | Currently participating in any other interventional clinical study within 30 days. | | |
| 9 | Patients who are considered not suitable for the study according to the investigator's judgment for the patient's best interest | | |

| Screen No. | Subject Initials Placebo Run-in<br>Visit 2 |
|---|---|
| Date of visit:// | (dd/mmm/yyyy) |
| Investiga | ional Product Administration |
| Is investigational product dispens | ed to subject: Yes* No |
| All the eligible subjects will receive PL | ACEBO during the run-in period |
| Date of dispense:/ | / (dd/mmm/yyyy) |
| Number of dispensed: F | Pack |

| Screen No. Subject I | Initials | Random No. | Baseline<br>Visit 3 |
|---|---|---|---|
| Date of visit://_ | (d | ld/mmm/yyyy) | |
| Ph | ysical Ex | aminations | |
| Is the examination performed: | Yes 🗌 N | 0 | |
| Date of examination:/ | / | (dd/mmm/yy | уу) |
| | R | esult | Specify if abnormal or |
| Sites/System | Normal | Abnormal | not done |
| 1 General appearance | | | |
| 2 Head/ears/eyes/nose/throat | | | |
| 3 Mouth | | | |
| 4 Skin | | | |
| 5 Neck (including thyroid) | | | |
| 6 Lymph nodes | | | |
| 7 Spine | | | |
| 8 Cardiovascular system | | | |
| 9 Respiratory system | | | |
| 10 Gastro-intestinal system | | | |
| 11 Nervous system | | | |
| 12 Musculoskeletal system | | | |
| 13 Blood and blood forming organs | | | |
| 14 Mental status | | | |
| Other, specify: | | | |

| S R | age 10 |
|---|---|
| Vital Signs | |
| Is the assessment performed: Yes No | |
| Date of assessment:/ (dd/mmm/yyyy) | |
| Body temperature:°C | |
| Pulse rate: bpm | |
| Respiratory rate: times/ minute | |
| Seated Office Blood Pressure | |
| Is the assessment performed*: Yes No *: the subject's office BP will be measured at an air-conditioned room after around 30 minutes of resisting position using an electronic sphygmomanometer | st in the |
| Date of assessment:/ (dd/mmm/yyyy) | |
| Systolic Blood Pressure: Right arm: mmHg | Нg |
| Diastolic Blood Pressure: Right arm: mmHg | |
| Eligibility Confirmation and Randomization Does subject meet the criteria*: Yes No The arm with higher SBP value should be used to re-confirm the inclusion criteria #2. | |
| Does subject enter Yes Random No.: R randomization: BP measurement arm <sup>8</sup> : Left arm Right arm 8: Blood pressure measurements (including office BP and 24-ABPM) in the following visits should be made on the same arm the higher value at baseline. | -hour |
| No, please fill in completion of study page. | |
| Signature | |
| Investigator's signature: Date: | |

Random No.

Subject Initials

Screen No.

Baseline

|------------|------------------|------------|---------------------|
| Screen No. | Subject Initials | Random No. | Baseline<br>Visit 3 |

| Is the asse | Is the assessment performed: Yes No | | | | |
|---|---|---|---|---|---|
| Date of as | sessment:/_ | | (đd/mn | nm/yyyy) | |
| Time | SBP (mmHg) | DBP (mmHg) | Time | SBP (mmHg) | DBP (mmHg) |
| 06 : 00 | | | 16 : 00 | | |
| 06:30 | | | 16 : 30 | | |
| 07 : 00 | | | 17 : 00 | | |
| 07 : 30 | | <del></del> | 17 : 30 | | |
| 08 : 00 | | | 18 : 00 | | |
| 08 : 30 | | Publication I | 18 : 30 | | |
| 09 : 00 | | | 19:00 | | |
| 09:30 | | | _19 : 30 | | MANAGEM CONTROL SALES |
| 10 : 00 | | | 20 : 00 | | |
| 10 : 30 | | · | 20 : 30 | | |
| 11 : 00 | | | 21 : 00 | | |
| 11 : 30 | | | 21 : 30 | | |
| 12 : 00 | Process Processed A | | 22 : 00 | | |
| 12 : 30 | | | 23 : 00 | | |
| 13 : 00 | <u> </u> | | 24 : 00 | | |
| 13 : 30 | | | 01 : 00 | | |
| 14 : 00 | | | 02 : 00 | province described balances | |
| 14 : 30 | | | 03 : 00 | | |
| 15 : 00 | | | 04 : 00 | | |
| 15 : 30 | | <u> </u> | 05 : 00 | | |

| | | Biochemistry Tests | | |
|---|---|---|---|---|
| ls th | Is the test performed: Yes No | | | |
| Date | e of sample:/ | / (dd/mmm/yyyy | ·) | |
| | _ | | | Result |
| | Item | Value | Normal | Abnormal |
| 1 | Total bilirubin | | | ☐cs ☐ncs |
| 2 | Aspartate transaminase (AST) | | | □cs □ncs |
| 3 | Alanine transaminase<br>(ALT) | | | □cs □ncs |
| 4 | Alkaline phosphatase<br>(ALP) | | | □cs □ncs |
| 5 | Serum creatinine | | | cs ncs |
| 6 | Blood urea nitrogen<br>(BUN) | | | □cs □ncs |
| 7 | Uric acid | | | ☐cs ☐ncs |
| 8 | Triglyceride (TG) | | | ☐cs ☐ncs |
| 9 | Total cholesterol (T-Cho) | | | ☐cs ☐ncs |
| 10 | HDL-cholesterol (HDL-C) | | | ☐cs ☐ncs |
| 11 | LDL-cholesterol (LDL-C) | | | ☐cs ☐ncs |
| 12 | Glucose (A.C.) | | | ☐cs ☐ncs |
| 13 | Hba1c | | | ☐cs ☐ncs |
| 14 | Sodium (Na) | | | ☐cs ☐ncs |
| 15 | Potassium (K) | | | ☐cs ☐ncs |
| 16 | Chloride (CI) | | | ☐cs ☐ncs |

|------------|------------------|------------|---------------------|
| Screen No. | Subject Initials | Random No. | Baseline<br>Visit 3 |

| | Hematology Tests | | | |
|---|---|---|---|---|
| ls t | Is the test performed: Yes No | | | |
| Da | te of sample:/ | /(dd/mmm/yyy | y) | |
| | Result | | | |
| | Item | Value | Normal | Abnormal |
| 1 | Hemoglobin | | | ☐cs ☐ncs |
| 2 | Platelet | | | ☐cs ☐ncs |
| 3 | RBC | | | ☐cs ☐ncs |
| 4 | WBC | | | ☐cs ☐ncs |
| 5 | Neurophils | | | ☐cs ☐ncs |
| 6 | Eosinophils | | | ☐cs ☐ncs |
| 7 | Lymphocyte | | | ☐cs ☐ncs |
| 8 | Monocytes | | | □cs-□ncs- |
| 9 | Basophils | | | ☐cs ☐ncs |
| 1 | | | | |
| | | Urinalysis Tests | | |
| ls t | he test performed: 🔲 🗅 | Yes No | | |
| Dat | e of sample:/ | /(dd/mmm/yyy | y) | |
| | 140.00 | <b>V</b> -1 | Result | |
| ltem | | Value | Normal | Abnormal |
| 1 | WBC | | | ☐cs ☐ncs |
| 2 | RBC | | | ☐cs ☐ncs |
| 3 | PH | | | ☐cs ☐ncs |
| 4 | PROTEIN | | | □cs □ncs |

SUGAR

|---|---|---|
| Biomarkers | for Blood Vessel Infla | mmation or Damage |
| ls the test performed: | Yes No | |
| Date of sample:/_ | /(dd/mmm | n/yyyy) |
| Iten | 1 | Result |
| 1 high sensitivity C-rea | ctive protein (hsCRP) | |
| 2 creatine kinase (CK/6 | CPK) | |
| | Electrocardiogram | (ECG) |
| Is the examination perform | med: Yes No | |
| Date of examination: | _//(dd/ | mmm/yyyy) |
| Result: Normal . | Abnormal, NCS Abnorm | nal, CS |
| Abnormal Findings: | | |
| <u> </u> | | |
| Name of the state | | |
| Inv | estigational Product A | dministration<br> |
| Is investigational product | dispensed to subject: | Yes No |
| Date of dispense: | | _(dd/mmm/yyyy) |
| Number of disper | ised: Pack | |
| Is investigational product | retrieved from subject: | Yes No |
| Date of retrieved: | | (dd/mmm/yyyy) |
| Number of retriev | red: Pack | |
| Number of lost: _ | Pack | |
| Number of taken: | Pack | |

Baseline

| Screen No. | Subject Initials | Random No. | Dietary<br>Visit 4 |
|------------|------------------|------------|--------------------|

| Date | of | visit: | _/_ | _/_ | (dd/mmm/yyyy) |
|------|----|--------|-----|-----|---------------|
|------|----|--------|-----|-----|---------------|

| | Physical Examinations | | | |
|---|---|---|---|---|
| ls ti | Is the examination performed: Yes No | | | |
| Dat | e of examination:/ | | (dd/mmm/yy | ууу) |
| | Sitas/System | Re | sult | Specify if abnormal or |
| | Sites/System | Normal | Abnormal | not done |
| 1 | General appearance | | | |
| 2 | Head/ears/eyes/nose/throat | | | |
| 3 | Mouth | | | |
| 4 | Skin | | | |
| 5 | Neck (including thyroid) | | | |
| 6 | Lymph nodes | | | |
| 7 | Spine | | | |
| 8 | Cardiovascular system | | | |
| 9 | Respiratory system | | | |
| 10 | Gastro-intestinal system | | | |
| 11 | Nervous system | | | |
| 12 | Musculoskeletal system | | | |
| 13 | Blood and blood forming organs | | | |
| 14 | Mental status | | | |
| 15 | Other, specify: | | | |

| Sur | een No. | Subject | וווונומוס | Nanc | ioni No. | Visit 4 |
|---|---|---|---|---|---|---|
| | | | Vita | l Signs | | |
| Is the as | sessment per | formed: | Yes 🗌 | No | | |
| Date of a | assessment: _ | / | | (dd/ | mmm/yyyy) | |
| Body ter | mperature: | <u>_</u> °C | | <u></u> | | |
| Pulse ra | te: b | pm | | | | |
| Respirat | tory rate: | times/ | minute | | <u></u> | |
| | | | | Second Second Delivery | | |
| | | Seate | ed Office | Blood F | ressure | |
| *: the sub<br>sitting pos | ssessment per<br>ject's office BP v<br>sition using an ele<br>ame equipment | vill be measu | red at an air | -conditioned | room after aro<br>urements have | und 30 minutes of rest in the to be made on the same arm |
| Date of | assessment: | /_ | | (dd/ | mmm/yyyy) | |
| Systolic | Blood Pressu | re : | mmHg | J | | |
| Diastolic | Blood Pressi | ıre: | mmHg | ] | | |
| | | | | | S 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
| | | nvestiga | tional Pr | oduct A | dministrati<br>— | on |
| Is invest | tigational prod | uct <b>dispen</b> | sed to sub | ject: | Yes No | |
| | Date of disper | ise:/_ | | | (dd/mmm/y) | /уу) |
| | Number of dis | pensed: | Pad | ck | | |
| Is invest | tigational prod | uct retrieve | ed from su | bject: | Yes No | |
| | Date of retriev | ed:/_ | /_ | | (dd/mmm/yy | уу) |
| | Number of ret | rieved: | Pack | <b>S</b> | | |
| | Number of los | t: | Pack | | | |
| | Number of tak | en: | Pack | | | |

Dietary

| Screen No. | Subject Initials | Random No. | Dietary<br>Visit 5 |
|------------|------------------|------------|--------------------|

| Date | of | visit: | /_ | <u> </u> | (dd/mmm/yyyy) |
|------|----|--------|----|----------|---------------|
|------|----|--------|----|----------|---------------|

| | Physical Examinations | | | |
|---|---|---|---|---|
| ls t | he examination performed: | Yes No | | |
| Daf | te of examination:/ | _/ | (dd/mmm/y <sub>)</sub> | ууу) |
| | 01410:4 | Re | sult | Specify if abnormal or |
| [<br> | Sites/System | Normal | Abnormal | not done |
| 1 | General appearance | | | |
| 2 | Head/ears/eyes/nose/throat | | | |
| 3 | Mouth | | | |
| 4 | Skin | | | |
| 5 | Neck (including thyroid) | | | |
| 6 | Lymph nodes | | | |
| 7 | Spine | | | |
| 8 | Cardiovascular system | | | |
| 9 | Respiratory system | | | |
| 10 | Gastro-intestinal system | | | |
| 11 | Nervous system | Victoria de la constanta de la | | |
| 12 | Musculoskeletal system | | | |
| 13 | Blood and blood forming organs | | | |
| 14 | Mental status | | | |
| 15 | Other, specify: | | | |

| Screen No. | Subject Initials | Random No. | Dietary<br>Visit 5 |
|------------|------------------|------------|--------------------|

| Vital Signs |
|---|
| Is the assessment performed: Yes No |
| Date of assessment:/ (dd/mmm/yyyy) |
| Body temperature:°C |
| Pulse rate: bpm |
| Respiratory rate: times/ minute |
| Seated Office Blood Pressure |
| Is the assessment performed*: Yes No *: the subject's office BP will be measured at an air-conditioned room after around 30 minutes of rest in the sitting position using an electronic sphygmomanometer. All measurements have to be made on the same arm and the same equipment |
| Date of assessment://(dd/mmm/yyyy) |
| _Systolic Blood Pressure : mmHg |
| Diastolic Blood Pressure: mmHg |
| Investigational Product Administration |
| Is investigational product <b>dispensed</b> to subject: Yes No |
| Date of dispense://(dd/mmm/yyyy) |
| Number of dispensed: Pack |
| Is investigational product <b>retrieved</b> from subject: Yes No |
| Date of retrieved://(dd/mmm/yyyy) |
| Number of retrieved: Pack |
| Number of lost: Pack |
| Number of taken: Pack |

| Screen No. | Subject Initials | Random No. | Dietary<br>Visit 6 |
|----------------|------------------|---------------|--------------------|
| Date of visit: | <u></u> | (dd/mmm/yyyy) | |

| | Physical Examinations | | | |
|---|---|---|---|---|
| ls ti | he examination performed: | Yes No | | |
| Dat | e of examination:/ | _/ | (dd/mmm/y) | ууу) |
| | 014101 | Re | sult | Specify if abnormal or |
| | Sites/System | Normal | Abnormal | not done |
| 1 | General appearance | | | |
| 2 | Head/ears/eyes/nose/throat | | | |
| 3 | Mouth | | | |
| 4 | Skin | | | |
| 5 | Neck (including thyroid) | | | |
| 6 | Lymph nodes | | | |
| 7 | Spine | | | |
| 8 | Cardiovascular system | | | |
| 9 | Respiratory system | | | |
| 10 | Gastro-intestinal system | | | |
| 11 | Nervous system | | | |
| 12 | Musculoskeletal system | | | |
| 13 | Blood and blood forming organs | | | |
| 14 | Mental status | | | |
| 15 | Other, specify: | | | |

| Vital Signs | |
|---|---|
| Is the assessment performed*: | |
| Date of assessment:/ /(dd/mmm/yyyy) | |
| Body temperature:°C | |
| Pulse rate: bpm | |
| Respiratory rate: times/ minute | |
| Seated Office Blood Pressure | |
| Is the assessment performed*: Yes No | |
| the subject's office BP will be measured at an air-conditioned room after around 30 minutes of rest in sitting position using an electronic sphygmomanometer. All measurements have to be made on the same and the same equipment | the<br>arm |
| Date of assessment:/(dd/mmm/yyyy) | |
| Systolic Blood Pressure : mmHg | |
| Diastolic Blood Pressure: mmHg | |

|------------|------------------|------------|--------------------|
| Screen No. | Subject Initials | Random No. | Dietary<br>Visit 6 |

| | 24 | 4-hour Ambula | itory SBI | P/DBP | |
|---|---|---|---|---|---|
| Is the asse | essment performed | : Yes N | 0 | | |
| Date of as | ssessment:/_ | | (dd/mn | nm/yyyy) | |
| Time | SBP (mmHg) | DBP (mmHg) | Time | SBP (mmHg) | DBP (mmHg) |
| 06 : 00 | | errennen Additional a | 16 : 00 | | |
| 06:30 | | | 16 : 30 | - | |
| 07 : 00 | | | 17 : 00 | | *************************************** |
| 07 : 30 | | | 17 : 30 | | |
| 08 : 00 | | | 18 : 00 | | |
| 08 : 30 | - | | 18 : 30 | | |
| 09 : 00 | | | 19 : 00 | | |
| 09 : 30 | | | 19 : 30 | | |
| 10 : 00 | | | 20 : 00 | | |
| 10 : 30 | | | 20 : 30 | | |
| 11:00 | | | 21 : 00 | · · <u></u> | |
| 11 : 30 | | | 21 : 30 | | |
| 12 : 00 | | | 22 : 00 | | |
| 12 : 30 | | | 23 : 00 | | |
| 13 : 00 | | | 24 : 00 | | |
| 13 : 30 | | | 01 : 00 | | |
| 14 : 00 | | | 02 : 00 | <u> </u> | |
| 14 : 30 | | | 03 : 00 | | |
| 15 : 00 | | | 04 : 00 | | |
| 15 : 30 | | | 05 : 00 | | |

|------------|------------------|------------|--------------------|
| Screen No. | Subject Initials | Random No. | Dietary<br>Visit 6 |

| | | Biochemistry Tests | Land Control | |
|---|---|---|---|---|
| ls th | ne test performed: Yes | ☐ No | | |
| Date | e of sample:/ | / (dd/mmm/yyyy | ') | |
| | | | | Result |
| | ltem | Value | Normal | Abnormal |
| 1 | Total bilirubin | | | ☐cs ☐ncs |
| 2 | Aspartate transaminase<br>(AST) | | | □cs □ncs |
| 3 | Alanine transaminase<br>(ALT) | | | □cs □ncs |
| 4 | Alkaline phosphatase<br>(ALP) | | | □cs □ncs |
| 5 | Serum creatinine | | | □cs □ncs |
| 6 | Blood urea nitrogen<br>(BUN) | | | □cs □ncs |
| 7 | Uric acid | | | □cs □ncs |
| 8 | Triglyceride (TG) | | | ☐cs ☐ncs |
| 9 | Total cholesterol (T-Cho) | | | CS NCS |
| 10 | HDL-cholesterol (HDL-C) | | | ☐cs ☐ncs |
| 11 | LDL-cholesterol (LDL-C) | | | csncs |
| 12 | Glucose (A.C.) | | | ☐cs ☐ncs |
| 13 | Hba1c | | | ☐cs ☐ncs |
| 14 | Sodium (Na) | | | ☐cs ☐ncs |
| 15 | Potassium (K) | | | ☐cs ☐ncs |
| 16 | Chloride (CI) | | | ☐cs ☐ncs |

| | | | | Visit 6 |
|---|---|---|---|---|
| S | S | R | | Page 23 |
| | | Hematology Tests | | |
| ls t | he test performed: Ye | es No | | |
| Da | te of sample:/ | / (dd/mmm/yyy | y) | |
| | Item | Value | | Result |
| | Item | value | Normal | Abnormal |
| 1 | Hemoglobin | | | ☐cs ☐ncs |
| 2 | Platelet | | | ☐cs ☐ncs |
| 3 | RBC | | | ☐cs ☐ncs |
| 4 | WBC | | | ☐cs ☐ncs |
| 5 | Neurophils | | | ☐cs ☐ncs |
| 6 | Eosinophils | | | ☐cs ☐ncs |
| 7_ | Lymphocyte | | | ☐cs ☐ncs |
| 8 | Monocytes | | | ☐cs ☐ncs |
| 9 | Basophils | | | ☐cs ☐ncs |
| | | | ; · | |
| | | Urinalysis Tests | | |
| ls t | he test performed: 🔲 Ye | es 🗌 No | | |
| Da | te of sample:/ | /(dd/mmm/yyy | y) | |
| | 140 | V-1 | | Result |
| | Item | Value | Normal | Abnormal |
| 1 | WBC | | | ☐cs ☐ncs |
| 2 | RBC | | | ☐cs ☐ncs |
| 3 | PH | | | ☐cs ☐ncs |
| 1 | PROTEIN | | | |

Dietary

cs

NCS

**SUGAR** 

| | Screen No. | Subject Initials | Random No. | Dietary<br>Visit 6 |
|---|---|---|---|---|
| | Piemen | rara for Blood Vos | sel Inflammation o | or Damage |
| lo 4 | | Yes No | ser milamination ( | or Damage |
| | | | (dd/mmm/yyyy) | |
| Dai | | | | esult |
| | | em | N | esuit |
| 1 | high sensitivity (<br>(hsCRP) | -reactive protein | | |
| 2 | creatine kinase | (CK/CPK) | | |
| | <u> </u> | | | |
| | | Electrocard | diogram (ECG) | |
| ls t | he examination pe | erformed: Yes | No | |
| Da | te of examination: | !! | (dd/mmm/yyyy) | |
| Re | sult: Normal | Abnormal, NCS [ | Abnormal, CS | |
| Abı | normal Findings: | | | |
| | | Investigational Pi | roduct Administrat | ion |
| ls i | nvestigational pro | duct <b>retrieved</b> from su | ubject: 🔲 Yes 📗 No | |
| | Date of retrie | ved://_ | (dd/mmm/y | ууу) |
| | | trieved: Pacl | | |
| | Number of lo | st: Pack | | |
| | Number of ta | ken: Pack | | |

|------------|---------------------------|------------------------------------|
| Screen No. | Subject Initials Random N | Follow-up o. Off-treatment Visit 7 |

| Date of visit: | _/ | _/ | (dd/mmm/yyyy |
|----------------|----|----|--------------|
|----------------|----|----|--------------|

| | Ph | ysical Exa | minations | |
|---|---|---|---|---|
| ls t | he examination performed: | Yes No | | |
| Dai | te of examination:/ | | (dd/mmm/y <sub>)</sub> | ууу) |
| | Sitos/Systom | Re | sult | Specify if abnormal or |
| | Sites/System | Normal | Abnormal | not done |
| 1 | General appearance | | | |
| 2 | Head/ears/eyes/nose/throat | | | |
| 3 | Mouth | | | |
| 4 | Skin | | | |
| 5 . | Neck (including thyroid) | | | |
| 6 | Lymph nodes | | | |
| 7 | Spine | | | |
| 8 | Cardiovascular system | | | |
| 9 | Respiratory system | | | |
| 10 | Gastro-intestinal system | | | |
| 11 | Nervous system | | | |
| 12 | Musculoskeletal system | | | |
| 13 | Blood and blood forming organs | | | |
| 14 | Mental status | | | |
| 15 | Other, specify: | | | |

| Vital Signs |
|---|
| Is the assessment performed: Yes No |
| Date of assessment://(dd/mmm/yyyy) |
| Body temperature:°C |
| Pulse rate: bpm |
| Respiratory rate: times/ minute |
| Seated Office Blood Pressure |
| Is the assessment performed*: Yes No |
| *: the subject's office BP will be measured at an air-conditioned room after around 30 minutes of rest in sitting position using an electronic sphygmomanometer. All measurements have to be made on the same a and the same equipment |
| Date of assessment:/(dd/mmm/yyyy) |
| Systolic Blood Pressure : mmHg |
| Diastolic Blood Pressure: mmHg |

| ।<br>\$ Investigational product; *: An AE that the outcome is death should be considered as a SAE | A | A | A | A | AE no.<br>Adverse Event | Is there any adverse event: Yes No Note: All the adverse events occurring from Baseline (Visit 3) to study completion (Visit 7)/withdrawal should be recorded. | | S | Screen No. |
|---|---|---|---|---|---|---|---|---|---|
| outcome is death should be considered | / | / | | | Onset Date<br>End date or Ongoing<br>(dd/mmm/yyyy) | is No Baseline (Visit 3) to study completion | Advers | | Subject Initials |
| as a SAE | | | | | Severity 1=Mild, 2=Moderate, 3=Severe | (Msit 7)/withdr | Adverse Event | <br> 70<br> | 73 |
| | | | l | | SAE<br>1= Yes,<br>2=No, | awal sho | | - Calculation | Random No. |
| Is this the I | _ | ] | | | Relationship to Study Drug 1=Certain, 2=Probable/Likely, 3=Possible, 4=Unlikely, 5=unrelated, 6=Unknown | ould be recorded. | | | No. |
| ls this the last page used? | | | | | Action Taken 1=IP <sup>\$</sup> not changed, , 2=IP interrupted, 3=IP withdrawn, | | | | |
| sed? 🔲 Yes | | | | l | Treatment Required 1=No, 2=Medication 3=Non-drug therapy, 4=Medication and non-drug therapy | | | Pag | |
| s No | | | <b>-</b> | <b> </b> | Outcome 1=Resolved 2=Persisting 3=Death* 4=Unknown | | | Page 27- ( ) | M Visit |

| Screen No. | 95 | Subject Initials | | Random No. | Ö | An Visit |
|---|---|---|---|---|---|---|
| S | | - Control of the Cont | | 22 | | Page 28- ( ) |
| | | Conc | comitant | Concomitant Medication | | |
| s there any concomitant medication: <br>lote: Antihypertensive medication or supplem | sation: Tes<br>supplements that the | No<br>the subjects too | k within 3 mo | nths prior to ICF date | will be recorded, All | s there any concomitant medication: 🔲 Yes 🦳 No<br>lote: Anthypertensive medication or supplements that the subjects took within 3 months prior to ICF date will be recorded. All the concomitant medication used from |
| Medication Medication Medication | Single dose | Unit a | Route b | Frequency c, | Indication <sup>d</sup> | Start Date End date or Ongoing |
| | | | | | | /or [ |
| | | | | | | /or |
| M | | | | | | |
| | | | | | | //or |
| ** MG ML, G, MCG, UG, TABLET, CAPSULE, DROPS 1=ORAL, 2=TOPICAL, 3=NASAL, 4=SUBLINGUAL, 5=INTRAVENOUS, 6=INTRAMUSCULAR, 7=INHALED, 8=SUBCUTANEOUS, 9=TRANSDERMAL, 10=OTHERS 10=OTHERS 11 OLD, T.I.D, B.I.D, Q12H, QD, HS, PRN, STAT 12 Please use the event code according to the AE page (A001~), Medical history page (H001~), or Prophylaxis/ routine (P000) | APSULE, DROPS,<br>4=SUBLINGUAL,<br>PRN, STAT | 5=INTRAVENC | NS, 6=INTR/ | MUSCULAR, 7=INF | HALED, 8=SUBCUTA | NEOUS, 9=TRANSDERMAL, |
| | | | | - PARENAMENTE | Is this the k | Is this the last page used? Yes No |

| Screen No. | Subject Initials | Random No. | Study Completion |
|------------|------------------|------------|------------------|

| End of Study/ Early Termination | |
|---|---|
| Date of the subject was taken off the study: | //(dd/mmm/yyyy) |
| Did the subject complete the study: | Yes No (If No, please record the primary reason) |
| Primary reason<br>for early<br>termination | <ul> <li>☐ Subject withdraw consent</li> <li>☐ Lost to follow up</li> <li>☐ Subjects who use prohibited medications, or any other</li> </ul> |
| | medications/therapies/supplements that could affect blood pressure Subjects stop taking investigational product, or temporarily interrupt |
| | taking investigational product over 1 week |
| | Protocol violation |
| | Pregnancy or lactating |
| | Subject with two value of blood pressure over the upper limit of stage I hypertension within one week, SBP ≥ 160 mmHg or DBP ≥ 100 mmHg |
| | Adverse event(s): |
| | Patients who are considered not suitable for the study according to the investigator's judgment for the patient's best interest |
| | Death, date of death:/(dd/mmm/yyyy) |
| | Other, please specify: |
| Comments: | |
| | Signature |
| | e report form have been entered under my authority and to the best of my curate and complete. |

Date:

Investigator's signature: